CLINICAL TRIAL: NCT07399600
Title: Personalized Transcranial Magnetic Stimulation for Metabolic Dysfunction and Alcohol-Related Liver Disease (MetALD): A Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Personalized Transcranial Magnetic Stimulation (TMS) for Metabolic Dysfunction and Alcohol-Related Liver Disease
Acronym: P-TMS MetALD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJP20250926
Record Dates: First submitted 2025-11-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Liver Diseases, Alcoholic; Fatty Liver; Metabolic Syndrome
Keywords: Liver Diseases, Alcoholic; Fatty Liver; Metabolic Syndrome; Transcranial Magnetic Stimulation; Randomized Controlled Trial
MeSH Terms: conditions — Liver Diseases, Alcoholic; Fatty Liver; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional rTMS (Active Comparator)
  Interventions: Device: Conventional rTMS
- Sham rTMS (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation Sham
- Active rTMS (Experimental)
  Interventions: Device: Individually Targeted rTMS

INTERVENTIONS:
Device: Individually Targeted rTMS — Participants will receive individualized transcranial magnetic stimulation (TMS) based on neuroimaging-guided localization of the nucleus accumbens (NAc). After the first MRI scan, participants will be randomized by an independent researcher responsible for data analysis. The individualized stimulation coordinates will be provided to the TMS operator before treatment.
  Intervention will be delivered using intermittent theta-burst stimulation (iTBS): the coil will be placed tangentially to the scalp over the individualized target. Stimulation parameters: 90% resting motor threshold (RMT); bursts of 3 pulses at 50 Hz; bursts repeated at 5 Hz; a total of 1800 pulses per session; stimulation duration 570 seconds. Each participant will receive 20 sessions in total, with at least 2 treatment days per week (2 sessions/day, 4 sessions/week). MRI and clinical assessments will be repeated at mid-treatment and after treatment completion, with follow-up clinical evaluations at 1, 3, and 6 months.
  Arms: Active rTMS
Device: Conventional rTMS — Conventional rTMS is applied to the left dorsolateral prefrontal cortex (DLPFC) using the standard 5 cm rule for scalp-based localization. Stimulation is delivered with intermittent theta-burst stimulation (iTBS) at 90% resting motor threshold (RMT), 3 pulses at 50 Hz per burst, repeated at 5 Hz, for a total of 1800 pulses per session. Each session lasts about 570 seconds. Participants complete 20 sessions over 4 weeks, with 2 sessions per day on 2 days per week.
  Arms: Conventional rTMS
Device: Transcranial Magnetic Stimulation Sham — Sham rTMS is delivered using a sham coil or low-intensity stimulation (10% RMT) to mimic the clicking sounds and scalp sensations of active rTMS without producing cortical activation. The sham sessions are matched to the active treatment in frequency, duration, and total number: 20 sessions in 4 weeks (2 sessions/day, 2 days/week, 570 seconds per session).
  Arms: Sham rTMS

SUMMARY:
The goal of this clinical trial is to learn if repetitive Transcranial Magnetic Stimulation (rTMS), a non-invasive brain stimulation technique, works to treat Metabolic dysfunction-associated and alcohol-associated liver disease (MetALD). The main questions it aims to answer are:

* Can rTMS effectively treat MetALD?
* Is an individualized, precision-targeted rTMS approach more effective than the standard rTMS method?
* What changes in brain activity are associated with the treatment?

Researchers will compare three different types of stimulation:

* Group A: Individualized rTMS targeting a deep brain reward area (the Nucleus Accumbens) based on each participant's brain scan (fMRI).
* Group B: Standard rTMS applied using the traditional "5 cm" rule for positioning.
* Group C: Sham (placebo) rTMS, which mimics the procedure but delivers no significant magnetic stimulation.

Participants will:

* Be randomly assigned to one of the three groups (A, B, or C).
* Undergo an MRI brain scan before starting treatment.
* Receive a total of 20 rTMS sessions, completing at least 4 sessions per week.
* Have additional MRI scans and clinical assessments halfway through and immediately after the treatment course.
* Attend follow-up visits at 1, 3, and 6 months after treatment completion to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to understand the study protocol, requirements, and restrictions, are fully informed of potential adverse events, are willing to comply with follow-up visits, and voluntarily sign the informed consent form before enrollment.
* Meet the diagnostic criteria for MASLD according to the Guidelines for the Prevention and Treatment of Metabolic (Non-Alcoholic) Fatty Liver Disease (2024 Edition), and fulfill the European definition of MetALD with moderate alcohol consumption (20-50 g/day for women; 30-60 g/day for men).
* Age between 18 and 65 years.
* Body mass index (BMI) > 24 kg/m².
* No history of alcohol abuse.

Exclusion Criteria:

* Contraindications to magnetic resonance imaging (MRI) or transcranial magnetic stimulation (TMS).
* Mild cognitive impairment, defined as Montreal Cognitive Assessment (MoCA) score < 25.
* Severe comorbid somatic diseases or neurological disorders.
* History of psychiatric disorders, or current use of antipsychotic medications.
* Pregnant or breastfeeding women, or those planning pregnancy.
* Previous TMS treatment within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Liver Fat Content (LFC) From Baseline to End of Treatment as Measured by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) | From baseline to the end of treatment (Week 4)

SECONDARY OUTCOMES:
Change in Controlled Attenuation Parameter (CAP, dB/m) From Baseline as Assessed by Vibration-Controlled Transient Elastography (FibroScan® VCTE) | From baseline to mid-treatment (Week 2), end of treatment (Week 4), and at 1-, 3-, and 6-month follow-up
Change in Liver Stiffness Measurement (LSM, kPa) From Baseline as Assessed by FibroScan® VCTE | From baseline to mid-treatment (Week 2), end of treatment (Week 4), and at 1-, 3-, and 6-month follow-up
LFC From Baseline as Measured by MRI-PDFF | From baseline to the end of treatment (Week 4)
Proportion of Participants Achieving ≥30% or ≥50% Reduction in LFC From Baseline | From baseline to the end of treatment (Week 4)
Change in Serum Levels of Liver Enzymes (ALT, AST, ALP, GGT [U/L]) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Serum Level of Albumin From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in International Normalized Ratio (INR) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Prothrombin Time (PT) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Serum Level of Total Bilirubin (TBIL) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Proportion of Participants With ALT Reduction >17 U/L From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Glucose Metabolism Markers (HOMA-IR [Index]; HOMA-β [Index]) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Glucose Metabolism Markers (HbA1c [%]) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Fasting Plasma Glucose (FPG) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Fasting Insulin From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Concentration of Conventional Lipid Panel (TC, TG, HDL-C, LDL-C, non-HDL-C, VLDL-C [mmol/L]) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Concentration of Apolipoproteins (Apo A1, Apo B [g/L]) From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Serum Lipoprotein(a) (Lp(a)) Concentration From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Serum Free Fatty Acids (FFA) Concentration From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Body Weight [kg] From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in BMI [kg/m²] From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Body Circumferences (Waist, Hip) [cm] From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Waist-to-Hip Ratio From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in General Food Craving Questionnaire-Trait (G-FCQ-T) Total Score From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
  G-FCQ-T The General Food Craving Questionnaire-Trait (G-FCQ-T) is a self-reported instrument used to assess the general tendency to experience food cravings. It comprises 21 items. Participants rate each item on a 6-point Likert scale ranging from 1 ("Never") to 6 ("Always"). The total score is the sum of all item ratings, with a possible range from 21 to 126. A higher total score indicates a more severe trait propensity for food craving.
Change in General Food Craving Questionnaire-State (G-FCQ-S) Total Score From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
  G-FCQ-S The General Food Craving Questionnaire-State (G-FCQ-S) is a self-reported instrument used to assess the current, momentary state of food craving. It comprises 15 items. Participants rate each item on a 6-point Likert scale ranging from 1 ("Strongly Disagree") to 6 ("Strongly Agree"). The total score is the sum of all item ratings, with a possible range from 15 to 90. A higher total score indicates a more intense current state of food craving.
Change in Score on Visual Analogue Scale (VAS) for Subjective Food Craving From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
  Subjective food craving is assessed using a Visual Analogue Scale (VAS). Participants indicate their current, momentary level of food craving by marking a point on a 100-mm horizontal line. The left endpoint (0 mm) is labeled "No food craving at all," and the right endpoint (100 mm) is labeled "The most intense food craving imaginable." The score is determined by measuring the distance from the left endpoint to the participant's mark, ranging from 0 to 100. A higher score indicates a more intense subjective feeling of food craving.
Change in Caloric intake recorded by the Mint Health App From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
Change in Alcohol Use Disorders Identification Test (AUDIT) Score From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
  The Alcohol Use Disorders Identification Test (AUDIT) is a simple, self-reported screening tool developed by the World Health Organization (WHO) to identify hazardous and harmful patterns of alcohol consumption. The questionnaire consists of 10 items. The first 8 items are scored on a scale from 0 to 4. Items 9 and 10 are scored 0, 2, or 4. The total score is the sum of all item ratings, with a possible range from 0 to 40. A higher total score indicates a greater likelihood of hazardous and harmful alcohol use, as well as possible alcohol dependence.
Change in Penn Alcohol Craving Scale (PACS) Score From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
  The Penn Alcohol Craving Scale (PACS) is a self-reported questionnaire designed to measure the intensity of an individual's craving for alcohol over the past week. The scale consists of 5 items assessing the frequency, duration, and intensity of craving, the ability to resist drinking, and the overall rating of craving. Each item is rated on a 6-point scale from 0 to 6, with varying verbal anchors for each item (e.g., "Never" to "Nearly All the Time"). The total score is the sum of all 5 item ratings, with a possible range from 0 to 30. A higher total score indicates a more severe level of subjective alcohol craving.
Change in Alcohol Consumption Assessed by the Timeline Followback (TLFB) Method From Baseline | baseline, mid-treatment (Week 2), end of treatment (Week 4), 1, 3, 6 months
  Alcohol consumption is assessed using the Timeline Followback (TLFB) method, a structured interview that provides a quantitative estimate of an individual's daily drinking. Using a calendar to aid recall, participants retrospectively report their daily alcohol consumption over a specified period (e.g., the past 30 days). The data is used to calculate key metrics such as the number of drinking days, the number of heavy drinking days, and the average number of standard drinks consumed per day or per week. A higher value indicates a greater level of alcohol consumption.

OTHER OUTCOMES:
Resting-State Functional Connectivity (rs-FC) Measured by fMRI | From baseline to mid-treatment (Week 2) and end of treatment (Week 4)
  Resting-state functional connectivity (rs-FC) will be assessed using functional magnetic resonance imaging (fMRI). This measures the temporal correlation of spontaneous brain activity between different neural regions, forming functional networks (e.g., Default Mode Network, Executive Control Network). The strength of connectivity is represented by correlation coefficients (z-values). A higher absolute value indicates stronger functional connectivity.
Amplitude of Low-Frequency Fluctuations (ALFF) Measured by fMRI | From baseline to mid-treatment (Week 2) and end of treatment (Week 4)
  The amplitude of low-frequency fluctuations (ALFF) will be calculated from resting-state fMRI data. It measures the intensity of spontaneous neural activity in specific brain regions. The value is typically presented as a normalized Z-score. A higher ALFF value indicates greater regional spontaneous neural activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang, China